CLINICAL TRIAL: NCT02858765
Title: Influence of Light on Sleep, Awakening, Electroencephalogram (EEG) and Cognitive Performances, and Medical Technology Assessment for Registration and Long-term EEG Analysis
Brief Title: Influence of Light on Sleep, Awakening, Electroencephalogram (EEG) and Cognitive Performances
Acronym: CHRONOSOMNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6187
Record Dates: First submitted 2016-05-30; First posted 2016-08-08 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Human Sleep and Chronobiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- white polychromatic light A (Experimental)
  Interventions: Other: Application of white polychromatic light for 2h30 at different times of day
- white polychromatic light B (Experimental)
  Interventions: Other: Application of white polychromatic light for 2h30 at different times of day
- white polychromatic light C (Experimental)
  Interventions: Other: Application of white polychromatic light for 2h30 at different times of day
- white polychromatic light D (Experimental)
  Interventions: Other: Application of white polychromatic light for 2h30 at different times of day

INTERVENTIONS:
Other: Application of white polychromatic light for 2h30 at different times of day

SUMMARY:
The purpose of this project is to study the influence of light on sleep, wakefulness, EEG activity and cognitive performances. The study aim also to evaluate techniques for registration and analysis of the EEG over periods of time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 to 40 years
* With a hint of Bodymass index (BMI) between 17 and 30 kg.m - 2
* Healthy subject determined by a clinical examination, a psychological interview, a blood test, a urine analysis and an ophthalmologic examination
* Topic Subject with a score <6 questionnaire PSQI ("Sleep Questionnaire Pittsburgh")
* Subject agreeing to maintain a regular sleep/wake rhythm during the study
* Subject agreeing to refrain from caffeine, nicotine, alcohol, psychotropic drugs, cannabis or other drugs during the study
* Signed informed consent
* Subject affiliated to a social protection scheme

Exclusion Criteria:

* somatic diseases: cardiovascular, respiratory, gastrointestinal, hematopoietic, Visual
* immune system diseases
* kidneys and urinary tract diseases
* endocrine and metabolic diseases
* neurological diseases
* infectious diseases
* thrombocytopenia or other malfunction of blood platelets
* Subject with risk of thrombosis, including subject with a history of phlebitis, smoker under oral contraceptive...
* Subject with an addiction to caffeine, nicotine, alcohol, psychotropic drugs, cannabis, or any other drug
* Subject treatment contraindicated or inadvisable in combination with heparin
* Allergy to neoprene or lycra
* Dysfunction of the temporomandibular joint (TMJD)
* Blood donation in the previous 3 months before the inclusion
* Participation in other clinical trials in the previous 3 months before the inclusion
* Work by shifts in the year preceding the inclusion
* Trans-meridian travel (> 2 time zones) in the month previous the inclusion
* Contraindications to the use of the medical device
* Impossibility to give enlightened information (subject in an emergency situation, understanding difficulties,...)
* Subject under safeguard of justice
* Subject under tutorship or curatorship
* Pregnancy (women of childbearing age)
* Breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Analysis of EEG activity | up to 56 hours
  sleep fragmentation
Cognitive performances assessed using Psychomotor vigilance task (PVT) | up to 56 hours
  Psychomotor vigilance task (PVT)
Cognitive performances assessed using Sustained Attention to Response Task (SART) | up to 56 hours
  Sustained Attention to Response Task (SART)
Cognitive performances assessed using Digit Symbol Substitution Test (DSST) | up to 56 hours
  Digit Symbol Substitution Test (DSST)
Cognitive performances assessed using N-back tasks | up to 56 hours
  N-back tasks
Cognitive performances assessed using Paced Visual Serial Addition Task (PVSAT) | up to 56 hours
  Paced Visual Serial Addition Task (PVSAT)
Cognitive performances assessed using Visual analogue scales (VAS) for motivation | up to 56 hours
  Visual analogue scales (VAS) for motivation
Cognitive performances assessed using Positive and Negative Affect Scale (PANAS) | up to 56 hours
  Positive and Negative Affect Scale (PANAS)
Cognitive performances assessed using Karolinska Sleepiness Scale (KSS) | up to 56 hours
  Karolinska Sleepiness Scale (KSS)
Cognitive performances assessed using Visual Comfort Scale (VCS) | up to 56 hours
  Visual Comfort Scale (VCS)
Cognitive performances assessed using Racing and Crowded Thoughts Questionnaire (RCTQ) | up to 56 hours
  Racing and Crowded Thoughts Questionnaire (RCTQ)
Cognitive performances assessed using Mental Effort Rating Scale (RSME) | up to 56 hours
  Mental Effort Rating Scale (RSME)
Cognitive performances assessed using Karolinska Drowsiness Test (KDT) | up to 56 hours
  Karolinska Drowsiness Test (KDT)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Glacet R, Reynaud E, Robin-Choteau L, Reix N, Hugueny L, Ruppert E, Geoffroy PA, Kilic-Huck U, Comtet H, Bourgin P. A comparison of four methods to estimate dim light melatonin onset: a repeatability and agreement study. Chronobiol Int. 2023 Feb;40(2):123-131. doi: 10.1080/07420528.2022.2150554. Epub 2022 Dec 15. PMID 36519316